CLINICAL TRIAL: NCT01185990
Title: Moderate to Severe Tinnitus as Measured by MEG and the Synchronous Neural Interaction™ Test: Template Development Study
Brief Title: Tinnitus Measured by MEG and Synchronous Neural Interaction™ Test: Template Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Orasi Medical, Inc. (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Todd Verdoorn, PhD, Chief Scientific Officer, Orasi Medical, Inc.
Other Study IDs: TTD 10 - 01
Record Dates: First submitted 2010-08-17; First posted 2010-08-20 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tinnitus subjects: Subjects with chronic, moderate to severe unilateral tinnitus.
- Healthy control subjects

SUMMARY:
The study is designed to identify specific patterns of brain functional activity associated with chronic, moderate to severe tinnitus through the use of resting-state MEG scans. Robust patterns identified in this study will be used as a biomarker for subsequent clinical evaluation of experimental drug treatments for tinnitus. This study will conduct MEG scans on approximately 30 to 75 subjects with tinnitus and approximately 15 healthy control subjects. MEG scans will be obtained for each subject following screening, clinical and tinnitus evaluations. A subset of 6 subjects from the tinnitus cohort will be invited to undergo evoked auditory assessment during an extended MEG scan session to identify cortical regions that respond to the auditory stimulus. These six subjects also will be evaluated with a single structural MRI scan to support high-resolution mapping of the localized cortical regions. MEG data will be analyzed to identify patterns of brain activity that are specifically associated with the presence of tinnitus using both standard approaches and the Orasi Synchronous Neural Interaction™ (SNI) test. MEG scan results also will be evaluated to identify specific patterns of functional activity that correlate with other measures of tinnitus severity such as the Iowa Tinnitus Handicap Scale. This study will test the hypothesis that moderate to severe tinnitus is associated with altered patterns of brain functional activity measured by a brief, resting-state MEG scan. This hypothesis will be tested by comparing resting-state MEG scans of tinnitus patients with those the of healthy control subjects collected during this study and available in Orasi's existing MEG scan database.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 75 years of age at the time of screening.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
* Subject is a non-smoker.
* Subject is judged to be in good health based on medical history and brief physical examination.
* Subject has a diagnosis of chronic, moderate to severe (Tinnitus Handicap Inventory score range of 38 - 76, inclusive), unilateral tinnitus of unknown etiology, or is participating in the study as a healthy control subject.

Exclusion Criteria:

* Subject has severe hearing impairment, external or middle ear diseases or temporomandibular joint disorders.
* Subject has a diagnosis of a significant neurological condition including Alzheimer's disease, Parkinson's disease, vascular dementia, Lewy body dementia or frontal temporal dementia, human immunodeficiency virus, multiple sclerosis, or severe traumatic brain injury.
* Subject has a history of primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder, delusional disorder) or bipolar disorder.
* Subject has a history of seizures, epilepsy, stroke, peripheral neuropathy, head trauma with persistent post-concussive symptoms, ADHD, dyslexia or other clinically significant neurological disease or cognitive impairment.
* Subject has a current episode of major depressive disorder.
* Subject has used antidepressants, anxiolytics, antipsychotics or antiepileptic medications in the past 6 months.
* Subject has a recent (within 2 years) history of alcohol or substance abuse/dependence.
* Subject has completed an MRI within 2 weeks prior to the MEG scan.
* Subject has metal braces or pacemaker that may interfere with the MEG scan.
* Subject is unable to complete the MEG scan procedure.
* The investigator has any concern regarding the safe participation of a subject in the study, or if for any other reason the investigator considers the subject inappropriate for study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic, moderate to severe unilateral tinnitus
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Correlated brain activity | 1 day
  MEG scan data will be analyzed using standard frequency domain approaches and the Orasi SNI test for correlated, synchronous activity.

SECONDARY OUTCOMES:
Tinnitus Severity Ratings | Up to 14 days
  The degree of tinnitus severity also will be evaluated using the Iowa Tinnitus Handicap Questionnaire (THQ), Tinnitus Handicap Inventory (THI) and a Visual Analog Scale (VAS) of Tinnitus Severity.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Golden, MD, Principal Investigator — Noran Neurological Clinic; Tami Helmer, MD, Principal Investigator — Radiant Research
Locations (2):
- United States (2):
  - Noran Neurological Clinic, Minneapolis, Minnesota
  - Radiant Research, Minneapolis, Minnesota